CLINICAL TRIAL: NCT00971191
Title: A Presurgical Study To Evaluate Molecular Changes That Occur In Human Non-Small Cell Lung Cancer Tissue After Short Term Exposure To PF-00299804
Brief Title: A Study In Patients Who Will Undergo Surgical Removal Of Non-Small Cell Lung Cancer To Evaluate Molecular Changes That Occur In Tumor Tissue After Short Term Exposure To PF-00299804
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A7471031
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Stage I - III surgical resection molecular change brief pre-operative exposure
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): Patients treated with brief exposure to PF-00299804 prior to surgical resection
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — Brief exposure (5- 11 days) to study drug prior to surgical resection

SUMMARY:
This study will enroll patients who are planned to undergo surgical removal of their tumor. The goal of the study is to evaluate the changes that occur in the tumor after brief (about 8 days) exposure to the study drug.

DETAILED DESCRIPTION:
The A7471031 study was terminated on May 2, 2012. The decision for unplanned study termination was triggered by feasibility of further conduct of this trial as only 22 of the protocol-specified 75 patients were enrolled since the study initiated in February 2010. Based on this low accrual rate it was determined that the study was highly unlikely to complete accrual and provide meaningful data. The discontinuation of the study is not due to any safety issue.

ELIGIBILITY:
Inclusion Criteria:

* Radiographs consistent with lung cancer for which resection is indicated upon histologic confirmation of non-small cell lung cancer.
* Patient willing to take PF-00299804 for 5 to 11 days and provide blood and tissue specimens as required in the study.

Exclusion Criteria:

* Prior or concurrent systemic anticancer therapy for cancer (immunotherapy, hormonotherapy, biological therapy, or chemotherapy) less than one year from time of consent.
* Prior or concurrent radiation therapy to tumor at site of planned resection.
* Congestive heart failure (LVEF < 50%), uncontrolled hypertension, significant ventricular arrythmia.
* Drugs that are highly dependent on CYP2D6 for metabolism, or are generally accepted to have a risk of causing Torsades de Pointes.
* Prior or concurrent radiation therapy to tumor at site of planned resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-02; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To identify the molecular changes which occur in human non-small cell lung cancer tissue after short-term exposure to PF-00299804 administered at 45 mg daily after a loading dose | 30 months

SECONDARY OUTCOMES:
To correlate molecular changes with specific gene and protein changes (eg, mutations, amplifications, over expression) in members of the EGFR and HER2 signal transduction pathways (eg, KRAS, EGFR, HER2) | 30 months
To assess the effect of short term treatment of PF-00299804 on serum levels of the extracellular domain of EGFR and other serum markers of HER signaling (eg, serum HER2/neu and serum E-cadherin) | 30 months
To assess the relationship between the pharmacokinetic parameters with molecular changes detected in non-small cell lung cancer | 30 months
To assess the safety and tolerability of PF-00299804 in this setting | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Los Angeles, California

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471031&StudyName=A%20Study%20In%20Patients%20Who%20Will%20Undergo%20Surgical%20Removal%20Of%20%20Non-Small%20Cell%20Lung%20Cancer%20To%20Evaluate%20Molecular%20Changes%20That%20Occur%20In%20T